CLINICAL TRIAL: NCT06690294
Title: Assessing the Impact of Perceptions of Unpredictability on Objective Measures of Food Consumption and Metabolism: A Natural History Study
Brief Title: Assessing the Impact of Perceptions of Unpredictability on Objective Measures of Food Consumption and Metabolism
Status: Not yet recruiting | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001980; 001980-DK
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-20

CONDITIONS: Healthy Volunteer; Obestity
Keywords: Healthy Volunteer; Obesity; Eating Behavior
MeSH Terms: conditions — Obesity; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteer: adults, age 18-60 years

SUMMARY:
Background:

Many people in the United States are overweight or obese. This natural history study will look into how life events during childhood can impact eating behaviors and weight gain as adults.

Objective:

To explore how childhood experiences affect adult eating behaviors.

Eligibility:

Healthy people aged 18 to 60 years.

Design:

Participants will have 3 clinic visits.

They will be screened with blood tests. They will answer questions about their alcohol and tobacco use.

At the next visit, participants will undergo these activities:

Parts of their body (such as waist, neck, and thighs) will be measured with a tape.

They will have an imaging scan to find out how much body fat they have.

They will start wearing a device like a wristwatch that measures their physical activity. They will wear this device for up to 10 days.

They will wear a device on their upper arm or belly that measures blood glucose (sugar) levels. Participants will wear this for 7-10 days.

They will answer questions about their education, childhood, and routines.

They will receive a kit to collect a stool sample at home.

At the last visit, participants will have these tests:

Participants will relax and breathe normally while wearing a clear, plastic canopy that fits over their entire head.

Blood samples will be taken before and after participants drink a sugary drink.

Participants will be offered a large selection of foods for lunch. They will eat as much as they want. Then they will answer questions about how they feel about food and themselves.

DETAILED DESCRIPTION:
Study Description:

The unpredictability schema - "a pervasive belief that other people cannot be trusted and future outcomes cannot be predicted or controlled" - has been hypothesized to (1) be shaped by parental/household dynamics and (2) impact appetitive and consumptive behaviors. However, studies on appetitive behaviors were mostly based on self-report and to our knowledge, no studies have examined objective measurements of energy intake or expenditure in association with unpredictability. Therefore, the current study seeks to examine whether the unpredictability schema as measured by a composite score of unpredictability assessments is associated with ad libitum food consumption and eating in the absence of hunger, measured objectively. Furthermore, we will examine the associations between the unpredictability schema and physical activity, resting metabolic rate/respiratory quotient, and glucose trajectories during an oral glucose tolerant test and continuous glucose monitoring in a cohort of healthy participants.

Objectives:

Primary Objective:

* To determine whether an association exists between unpredictability schema measures (schema/beliefs and childhood experiences as measured by derived from the Child Unpredictability Index, Scale of Unpredictability Beliefs, Unpredictability Schema Scale, and Confusion, Hubbub, and Order Scale and, individually, by scale totals and subscales) and ad libitum food intake.
* To determine whether an association exists between the unpredictability schema and experience scores and eating in the absence of hunger (as determined by the snack food taste test).

Secondary Objectives:

* To determine whether an association exists between measures of the unpredictability schema and experience scores and physical activity.
* To determine whether an association exists between measures of the unpredictability schema and experience scores and resting metabolic rate and RQ.
* To determine whether an association exists between measures of the unpredictability schema and experience scores and glucose values (CGM and OGTT).
* To determine whether an association exists between measures of the unpredictability schema and experience scores and telomere length.
* To determine whether an association exists between measures of the unpredictability schema and experience scores and with gut microbiota composition.

Tertiary Objectives:

* To determine the associations between measures of early childhood experiences (as measured by an overall composite measure derived by the maternal care/warmth subscale of the Parental Bonding Instrument and physical and emotional neglect subscales from the Childhood Trauma Questionnaire and, individually, by scale totals and subscales) and outcomes outlined in the primary and secondary objectives.
* To determine whether an association exists between measures of early childhood experiences and the unpredictability schema and experience scores.
* Examine psychosocial and physiological variables (based on theory and past literature) that may mediate or moderate the relationship between the unpredictability schema and our primary and secondary endpoints.
* Examine associations of metabolic measures with psychosocial measures (e.g., perceived stress, anhedonia, anxiety, depression, etc.), hormonal endpoints, or future biomarker assayed at a later time point.

Endpoints:

Primary Endpoint:

* Ad libitum Food Intake (kcal) measured from a buffet meal task.
* Eating in the absence of hunger (kcal) from a snack food taste test.

Secondary Endpoints:

* Physical activity values and trajectories from the 10-day outpatient actigraphy assessment.
* Resting metabolic rate and respiratory quotient values obtained from the metabolic hood.
* Glucose values and trajectories from fasting labs, OGTT, and 10-day outpatient CGM assessment.
* Telomere length (t/s ratio)
* Gut Flora Composition

Tertiary Endpoints:

* Ad libitum Food Intake (kcal) measured from (1) a buffet meal task and (2) the snack food taste test; Physical activity values and trajectories from the 10-day outpatient actigraphy assessment; Resting metabolic rate and respiratory quotient values obtained from the metabolic hood; Glucose values and trajectories from fasting labs, OGTT, and 10-day outpatient CGM assessment.
* Ad libitum Food Intake (kcal) measured from (1) a buffet meal task and (2) the snack food taste test; Physical activity values and trajectories from the 10-day outpatient actigraphy assessment; Resting metabolic rate and respiratory quotient values obtained from the metabolic hood; Glucose values and trajectories from fasting labs, OGTT, and 10-day outpatient CGM assessment.
* Unpredictability schema and experience scores
* Ad libitum Food Intake (kcal) measured from (1) a buffet meal task and (2) the snack food taste test; Physical activity values and trajectories from the 10-day outpatient actigraphy assessment; Resting metabolic rate and respiratory quotient values obtained from the metabolic hood; Glucose values and trajectories from fasting labs, OGTT, and 10-day outpatient CGM assessment.
* Plasma hormone, metabolite and protein concentration measured following data collection.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Stated willingness to comply with all study procedures and availability for the duration of the study.
* 18-60 years of age.
* Able to read and understand English proficiently (to be able to complete the multiple study questionnaires and instruments).

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Diabetes

  * Random glucose >= 200 mg/dl or HbA1c >= 6.5% or
  * Self-reported history of type 1 or type 2 diabetes.
* Endocrine disorders, such as

  --Self-reported history of Cushing's disease, pituitary disorders, or hypo- and hyperthyroidism
* TSH <0.1 or >= 10 uIU/mL
* Pulmonary disorders

  --Self-reported history of chronic obstructive pulmonary disease or other lung disease that which would limit ability to follow the protocol (investigator judgment)
* Cardiovascular diseases,

  --Self-reported history of coronary heart disease, heart failure, arrhythmias, and peripheral artery disease that which would limit ability to follow the protocol (investigator judgment)
* Liver disease,

  * Advanced liver disease (as determined by history, labs, exams, and patient self-report) that which would limit ability to follow the protocol (investigator judgment)
  * AST or ALT elevations > 3 times upper limit of normal
* Gastrointestinal Surgery

  --Self-reported history of bariatric surgery
* Renal disease

  * Self-reported history of renal replacement therapy
  * Abnormal kidney function (defined as eGFR <60 mL/min/1.73m^2) determined at screening (eGFR values are computed using the 2021 CKD-epi equation)
* Central nervous system disease:

  --Including self-reported history of previous history of cerebrovascular accidents, dementia, and neurodegenerative disorders
* Infectious disease:

  --Self-reported history of active tuberculosis, HIV, chronic coccidiomycosis or other chronic or acute infections
* For Females: pregnancy, <=6 months postpartum, currently breastfeeding, or on birth control (i.e., ingested, injected or implanted; non-hormonal methods such as copper IUD will be allowed)
* Measured weight: greater than or equal to 450 lb. (maximum weight allowed on the DXA scanning tables by the manufacturer)
* Inability to provide informed consent.
* Self-reported history of psychological conditions including (but not limited to), active psychosis, schizophrenia, eating disorders, or forms of mental incapacity that would be incompatible with safe and successful participation in this study.
* Current use of medications/dietary supplements/alternative therapies known to alter energy metabolism.
* Inability to consume provided food during ad libitum food intake or snack food test based on a food allergy or intolerances or diet restrictions.
* Any disorder not covered by any other exclusion criteria which, in the investigator's and/or team's opinion jeopardizes the safety of the participant or others or would interfere with adherence to the protocol.
* Alcohol Abuse as defined by >= 8-point score on the Alcohol Use Disorders Identification Test (AUDIT) questionnaire will be an exclusion criterion.
* Current use of tobacco products that exceed "Very Low Dependence" on the Fagerstrom Test for Nicotine Dependence Tool (score greater than 2) will be an exclusion criterion.

Non-English-speaking subjects as a population will be excluded from participation in this protocol. Primary and secondary hypotheses of the protocol relate to a battery of psychological questionnaires and performances tests which are administered throughout the study. There are currently no validated, translated forms of these questionnaires and tests available; therefore, we will restrict enrollment to English speaking subjects only.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study will enroll healthy, non-pregnant, women and men aged 18-60 years old who are without diabetes from the Greater Phoenix area, Arizona, United States. The study anticipates screening/enrolling 310 participants to achieve a goal of 110 participants completing the study.
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
To determine whether an association exists between unpredictability schema measures and ad libitum food intake. | Day 10
  Ad libitum Food Intake (kcal) measured from a buffet meal task.
To determine whether an association exists between the unpredictability schema and experience scores and eating in the absence of hunger | Day 10
  Eating in the absence of hunger (kcal) from a snack food taste test.

SECONDARY OUTCOMES:
To determine whether an association exists between measures of the unpredictability schema and experience scores and physical activity. | Day 10
  Physical activity values and trajectories from the 10-day outpatient actigraphy assessment
To determine whether an association exists between measures of the unpredictability schema and experience scores and resting metabolic rate and RQ. | Day 10
  Resting metabolic rate and respiratory quotient values obtained from the metabolic hood.
To determine whether an association exists between measures of the unpredictability schema and experience scores and glucose values (CGM and OGTT) | Day 10
  Glucose values and trajectories from fasting labs, OGTT, and 10-day outpatient CGM assessment, including mean, standard deviation, area-under-the-curve, and estimated a1c
To determine whether an association exists between measures of the unpredictability schema and experience scores and telomere length | Day 10
  Telomere length (t/s ratio)
To determine whether an association exists between measures of the unpredictability schema and experience scores and with gut microbiota composition. | Day 10
  Gut Flora Composition

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Cabeza De Baca, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institute of Diabetes and Digestive and Kidney Disorders (NIDDK), Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001980-DK.html